CLINICAL TRIAL: NCT06396988
Title: Clinical Efficacy of Calcium and Sodium Phosphosilicate (Novamin) in the Treatment of MIH (Molar Incisor Hypolimineralization) in Pediatric Patients: Randomized Clinical Trial
Brief Title: Clinical Efficacy of Calcium and Sodium Phosphosilicate (Novamin) in the Treatment of MIH (Molar Incisor Hypolimineralization) in Pediatric Patients
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-MIHNOVAMIN
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Intervention Model Description: Split-mouth study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Novamin (Experimental)
  Interventions: Other: Novamin application
- Parodontax (Active Comparator)
  Interventions: Other: Parodontax application

INTERVENTIONS:
Other: Novamin application — Teeth from this group will be treated with the application of Sensodyne Repair&Protect Toothpaste for 28 days after each visit (1 application per day for 2 minutes).
  Arms: Novamin
Other: Parodontax application — Teeth from this group will be treated with the application of Parodontax Complete Protection Toothpaste for 28 days after each visit (1 application per day for 2 minutes).
  Arms: Parodontax

SUMMARY:
The aim of the following study is to evaluate the clinical efficacy of a toothpaste with calcium and sodium phosphosilicate in the treatment of demineralization of the dental enamel of molars and incisors in pediatric patients. Patients who agree to participate to the study will use 2 different toothpaste Sensodyne Repair and Protect and Parodontax, which will used with split mouth design. The following indices will be measured: BEWE, Bleeding Index, Gingival Index, Plaque Index, Dental sensitivity test- Schiff, Pain Intensity Index- VAS and PPD.

DETAILED DESCRIPTION:
Informed consent will be signed by the parents of the patients underage and will be asked the approval for the attendance of the study. To the parents of pediatric patients will be given for free the 2 toothpastes and will be explain the correct procedures for home oral care. The method used in the study is "Split-Mouth" design, in which contralateral teeth with MIH will used for control group. For the study the patients must have at least two demineralizations present on contralateral permanent molars or incisors. The toothpaste used for the study consist in 2 different types: Sensodyne Repair&Protect (used for the Trial group) and Parodontax Complete Protection (used for the control group).

The 2 toothpastes will be applied once a day, before going to sleep after normal oral hygiene, for at least two minutes for 28 days after each meeting. The products must be used in minimal quantities, in pea-size doses, applying it on the tooth with the finger while performing a massage, under the supervision of the parents and then rinsing.

At each meeting will be taken all the indices and the timing is: T0- study begin, T1- after 1 month, T2-after 3 months, T3- after 6 months, T4- after 9 months, T5- after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 2 demineralizations of the dental enamel of molars and incisors (molar incisor hypomineralization-MIH) on contralateral permanent teeth
* Patients with mild or moderate MIH
* Good general health (absence of particular systemic pathologies)

Exclusion Criteria:

* Patients undergoing orthodontic therapy
* Patients taking drugs
* Patients with severe MIH (tooth surface with defect > 2/3, post-eruptive enamel breakage)

Ages: 7 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2027-01-10 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
Change in Bleeding Index | Study begin, 1, 3, 6, 9, 12 months
  0: absence of bleeding after 30 seconds
  1. bleeding observed after 30 seconds
  2. immediate bleeding
Change in Gingival Index | Study begin, 1, 3, 6, 9, 12 months
  0: normal gingiva
  1. mild inflammation, edema and swelling, no bleeding
  2. moderate inflammation with edema, sweelling and bleeding on probing
  3. severe inflammation with marked edema, redness tissues, ulceration and spontaneous bleeding
Change in Plaque Control Record | Study begin, 1, 3, 6, 9, 12 months
  The index is calculated multiplying the total number of surfaces with plaque per 100
Change in Schiff Air Index | Study begin, 1, 3, 6, 9, 12 months
  0: the subject did not respond to air blasting
  1. the subject responded to air blasting
  2. the subject responded to air blasting and requested discontinuation
  3. the subject responded to air blasting, requested discontinuation and considered the stimulus to be painful
Change in Basic Erosive Wear Examination | Study begin, 1, 3, 6, 9, 12 months
  0: no erosive tooth wear
  1. initial loss of surface texture
  2. distinct defect, hard tissue loss < 50% of the surface area
  3. hard tissue loss ≥ 50% of the surface area
Change in Wong- Backer faces pain rating scales | Study begin, 1, 3, 6, 9, 12 months
  0-1: no pain 1-2: milde pain 3-4: moderate pain 5-6: acute pain 7-8: very severe pain 9-10: unbearable pain

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, DDS, PhD, Principal Investigator — University of Pavia
Locations (1):
- Unit of Orthodontics and Pediatric Dentistry - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Pediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to the PI.